CLINICAL TRIAL: NCT05630846
Title: A Phase II, Single-blind, Randomized, Controlled Study to Evaluate the Immunogenicity and Safety of a Measles, Mumps, Rubella, Varicella Vaccine Compared With ProQuad, Administered in Healthy Children 4-6 Years of Age
Brief Title: A Study on the Immune Response and Safety of a Combined Measles, Mumps, Rubella, Chickenpox Vaccine Compared to a Marketed Combined Vaccine, Given to Healthy Children 4 to 6 Years of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 217715; 2022-501564-18 (EudraCT Number)
Record Dates: First submitted 2022-11-24; First posted 2022-11-30 (Actual); Results first posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Measles; Mumps; Rubella; Chickenpox; Measles
Keywords: Measles; Mumps; Rubella; Varicella
MeSH Terms: conditions — Measles; Mumps; Rubella; Chickenpox | interventions — measles, mumps, rubella, varicella vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Single-blind study. Recipients and care providers will be unaware of vaccine administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- MMRV(H)NS Group (Experimental): Participants receive a single dose of an investigational measles, mumps, and rubella (MMR) at release potency and varicella at high (V[H]NS) potency vaccine on Day 1.
  Interventions: Biological: Investigational MMRV(H)NS vaccine
- MM(H)RVNS Group (Experimental): Participants receive a single dose of an investigational measles, rubella (MR), and varicella (VNS) at release potency and mumps at high (M[H]) potency vaccine on Day 1.
  Interventions: Biological: Investigational MM(H)RVNS vaccine
- M(L)M(L)R(L)V(L)NS Group (Experimental): Participants receive a single dose of an investigational measles, mumps, rubella (MMR), and varicella (VNS), all at low (L) potency vaccine on Day 1.
  Interventions: Biological: Investigational M(L)M(L)R(L)V(L)NS vaccine
- MMRV_Lot 1 and Lot 2 Pooled Group (Active Comparator): Participants receive a single dose of a marketed measles, mumps, rubella (MMR), and varicella (V) vaccine of Lot 1 or of 1 vaccine dose of a marketed MMRV vaccine of Lot 2 on Day 1.
  Interventions: Biological: Marketed MMRV_Lot 1 and Lot 2 vaccine

INTERVENTIONS:
Biological: Investigational MMRV(H)NS vaccine — 1 dose of a measles, mumps, and rubella at release potency and VNS at high (H) potency vaccine administered subcutaneously.
  Arms: MMRV(H)NS Group
Biological: Investigational MM(H)RVNS vaccine — 1 dose of a measles, rubella, and varicella at release potency and mumps at high (H) potency vaccine administered subcutaneously.
  Arms: MM(H)RVNS Group
Biological: Investigational M(L)M(L)R(L)V(L)NS vaccine — 1 dose of measles, mumps, rubella, and varicella, all at low (L) potency vaccine administered subcutaneously.
  Arms: M(L)M(L)R(L)V(L)NS Group
Biological: Marketed MMRV_Lot 1 and Lot 2 vaccine — 1 dose of a marketed measles, mumps, rubella, and varicella of Lot 1 or 1 dose of a marketed measles, mumps, rubella, and varicella of Lot 2 vaccine administered subcutaneously.
  Other Names: ProQuad
  Arms: MMRV_Lot 1 and Lot 2 Pooled Group

SUMMARY:
The main purpose of this study is to assess immune response and safety of various potencies of a measles, mumps, rubella, and varicella (MMRVNS) vaccines given to healthy children of 4 to 6 years of age.

DETAILED DESCRIPTION:
This study is designed to evaluate the immunogenicity and safety of the investigational measles, mumps, rubella, varicella vaccine (referred to as the MMRVNS vaccine) compared with the licensed measles, mumps, rubella, varicella vaccine, ProQuad (referred to as the MMRV vaccine), when given as a second dose to children 4 to 6 years of age who were previously primed with a first dose of any combination of measles, mumps, rubella, and varicella-containing vaccine(s).

This study will evaluate immunogenicity and safety using 3 MMRVNS formulations which vary for some or all the individual virus potencies. The 3 MMRVNS formulations (designated as MMRV(H)NS vaccine, MM(H)RVNS vaccine and M(L)M(L)R(L)V(L)NS vaccine) will be compared with the MMRV vaccine. To ensure representative data on the comparator, participants enrolled in the MMRV group will be randomized to two different lots (designated as MMRV_Lot 1 and MMRV_Lot 2). Throughout the study, the two lots will be analyzed as a pooled group.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants as established by medical history and clinical examination before entering into the study.
* A male or female between, and including, 4 years and 6 years of age (i.e., from 4 year birthday until the day before the 7-year birthday) at the time of study intervention administration, and in accordance with local regulations.
* Participant who previously received a first dose of varicella-containing vaccine in the second year of life.
* Participant who previously received a single dose of measles-, mumps-, rubella-containing vaccine in the second year of life.
* Written informed consent obtained from the participants' parent(s)/legally acceptable representative(s) (LAR[s]) prior to performance of any study-specific procedure (participant informed assent will be obtained from participants in line with local rules and regulations).
* Participants' parent(s)/LAR(s), who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g., completion of electronic diaries [eDiaries], return for follow-up visits).

Exclusion Criteria:

Medical Conditions

* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study interventions including hypersensitivity to neomycin or gelatin.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Hypersensitivity to latex.
* Major congenital defects, as assessed by the investigator.
* History of measles, mumps, rubella, or varicella disease.
* Recurrent history of or uncontrolled neurological disorders or seizures.
* Acute disease at the time of enrollment. Acute disease is defined as the presence of a moderate or severe illness with or without fever. Fever is defined as body temperature >=38.0 degrees Celsius (°C) (100.4 degrees Fahrenheit [°F)] by any age-appropriate route. All study interventions can be administered to participants with a minor illness such as diarrhea, mild upper respiratory infection without fever.
* Participant with history of coronavirus disease 2019 (COVID-19) who is still symptomatic.
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.

Prior and Concomitant Therapy

* Use of any investigational or non-registered product (drug, vaccine, or medical device) other than the study interventions during the period beginning 30 days before the dose of study interventions (Day -29 to Day 1), or their planned use during the study period.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting 90 days prior to the study intervention administration. For corticosteroids, this will mean prednisone equivalent >= 0.5 mg/kg/day or 20 mg/day whichever is the maximum dose for pediatric participants. Inhaled and topical steroids are allowed.
* Administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting 180 days before the dose of study interventions or planned administration during the study period.
* Administration of long-acting immune-modifying drugs at any time during the study period (e.g., infliximab).
* Previous vaccination with a second dose of varicella-containing vaccine or measles-, mumps-, rubella-containing vaccine.
* Administration or planned administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the dose and ending at 43 days after the dose of study interventions administration* (Visit 3), with the exception of:

  * inactivated influenza (flu) vaccine which may be given at any time during the study and administered at a different location than the study interventions and,
  * routinely recommended licensed childhood DTPa-containing vaccines which can preferably be co-administered according to the local immunization practices of the participating country.
* Any other age-appropriate vaccine may be given starting at Visit 3 and anytime thereafter.

  * In case an emergency mass vaccination for an unforeseen public health threat (e.g., a pandemic) is recommended and/or organized by public health authorities outside the routine immunization program, the time period described above can be reduced if necessary for that vaccine, provided it is used according to the local government recommendations and that GSK/IQVIA is notified accordingly.

Prior/Concurrent Clinical Study Experience

• Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational intervention (drug/invasive medical device).

Other Exclusions

* Child in care.
* Any study personnel's immediate dependents, family, or household members.
* Participants with the following high-risk individuals in their household:

  * Immunocompromised individuals
  * Pregnant women without documented history of varicella.
  * Newborn infants of mothers without documented history of varicella.
  * Newborn infants born <28 weeks of gestation.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 801 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (40):
- United States (33):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Bellflower, California
  - GSK Investigational Site, Huntington Park, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, Roseville, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Jose, California
  - GSK Investigational Site, Santa Clara, California
  - GSK Investigational Site, West Covina, California
  - GSK Investigational Site, Miami Lakes, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Ammon, Idaho
  - GSK Investigational Site, Idaho Falls, Idaho
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Lafayette, Louisiana
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Bingham Farms, Michigan
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Simpsonville, South Carolina
  - GSK Investigational Site, Tullahoma, Tennessee
  - GSK Investigational Site, Dickinson, Texas
  - GSK Investigational Site, McAllen, Texas
  - GSK Investigational Site, Richmond, Texas
  - GSK Investigational Site, Layton, Utah
  - GSK Investigational Site, Provo, Utah
  - GSK Investigational Site, Roy, Utah
  - GSK Investigational Site, South Jordan, Utah
- Colombia (2):
  - GSK Investigational Site, Barranquilla
  - GSK Investigational Site, Bogotá
- GSK Investigational Site, Riga, Latvia
- GSK Investigational Site, San Juan, Puerto Rico
- Taiwan (3):
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of the 801 participants enrolled, 796 were included in the Exposed set and started the study.
Pre-assignment Details: The participants enrolled in the measles, mumps, rubella, and varicella vaccine (investigational vaccine) (MMRVNS) groups were randomized to 3 formulations which varied in some or all the individual viral potencies. Participants enrolled in the measles, mumps, rubella, and varicella vaccine (comparator vaccine) (MMRV) group were randomized to 2 different lots. Throughout the study, the 2 lots were analyzed as a pooled group.
Groups:
- MMRV(H)NS Vaccine: Participants received a single dose of measles,mumps, and rubella (MMR) at release potency and varicella at high (V[H]NS) potency vaccine on Day 1.
- MM(H)RVNS Vaccine: Participants received a single dose of measles,rubella (MR), and varicella (VNS) at release potency and mumps at high (M[H]) potency vaccine on Day 1.
- (MMRV)(L)NS Vaccine: Participants received a single dose of MMR and VNS, all at low (L) potency vaccine on Day 1.
- MMRV_Lot 1 and Lot 2 Pooled Group: Participants received a single dose of a marketed MMRV vaccine from Lot 1 or Lot 2 on Day 1.
Period: Overall Study
Arm/Group | MMRV(H)NS Vaccine | MM(H)RVNS Vaccine | (MMRV)(L)NS Vaccine | MMRV_Lot 1 and Lot 2 Pooled Group
Started | 198 | 200 | 203 | 195
Completed | 187 | 192 | 197 | 189
Not Completed | 11 | 8 | 6 | 6
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 3 | 4 | 1
Not completed — Lost to Follow-up | 6 | 5 | 2 | 5
Not completed — Other | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- MMRV(H)NS Vaccine: Participants received a singledose of MMRV(H)NS vaccine on Day1.
- MM(H)RVNS Vaccine: Participants received a single dose of MM(H)RVNS vaccine on Day 1.
- (MMRV)(L)NS Vaccine: Participants received a single dose of M(L)M(L)R(L)V(L)NS vaccine on Day 1.
- Total: Total of all reporting groups
Arm/Group | MMRV(H)NS Vaccine | MM(H)RVNS Vaccine | (MMRV)(L)NS Vaccine | MMRV_Lot 1 and Lot 2 Pooled Group | Total
Number analyzed (Participants) | 198 | 200 | 203 | 195 | 796
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at time of first vaccination.
  years | 4.2 (0.4) | 4.2 (0.5) | 4.2 (0.5) | 4.2 (0.5) | 4.2 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 85 | 105 | 99 | 362
  Male | 125 | 115 | 98 | 96 | 434
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 34 | 33 | 33 | 33 | 133
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 25 | 36 | 33 | 37 | 131
  White | 123 | 113 | 115 | 109 | 460
  More than one race | 15 | 17 | 19 | 15 | 66
  Unknown or Not Reported | 1 | 1 | 3 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: GMC of Anti-measles Antibodies at Day 43
Description: Anti-measles antibodies were measured with multiplex luminex based immuno assay and the results were expressed as GMC, in milli international units per milliliter (mIU/mL). Analysis was performed on per protocol set which included all eligible participants who received study intervention as per protocol, were not unblinded, had immunogenicity results pre- and post-dose for at least 1 antigen, complied with blood draw interval between study intervention and post- dose blood sample, without intercurrent medical conditions that may interfere with immunogenicity and without prohibited concomitant medication/vaccination. Only participants with data available at specified timepoint were included in the analysis.
Time Frame: At Day 43
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Groups:
- MMRV(H)NS Vaccine: Participants received a single dose of MMRV(H)NS vaccine on Day1.
Arm/Group | MMRV(H)NS Vaccine | MM(H)RVNS Vaccine | (MMRV)(L)NS Vaccine | MMRV_Lot 1 and Lot 2 Pooled Group
Number analyzed (Participants) | 167 | 171 | 162 | 168
mIU/mL | 801 (691) [691 to 928] | 788 (682) [682 to 910] | 728 (622) [622 to 852] | 682 (581) [581 to 801]

2. Primary Outcome: GMC of Anti-mumps Antibodies at Day 43
Description: Anti-mumps antibodies were measured with multiplex luminex based immuno assay and the results were expressed as GMC, in arbitrary units per milliliter (AU/mL). Analysis was performed on per protocol set. Only participants with data available at specified timepoint were included in the analysis.
Time Frame: At Day 43
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | MMRV(H)NS Vaccine | MM(H)RVNS Vaccine | (MMRV)(L)NS Vaccine | MMRV_Lot 1 and Lot 2 Pooled Group
Number analyzed (Participants) | 167 | 171 | 162 | 168
AU/mL | 3369 (2976) [2976 to 3814] | 4770 (4259) [4259 to 5342] | 3114 (2771) [2771 to 3499] | 3176 (2830) [2830 to 3563]

3. Primary Outcome: GMC of Anti-rubella Antibodies at Day 43
Description: Anti-rubella antibodies were measured with multiplex luminex based immuno assay and the results were expressed as GMC, in international units per milliliter (IU/mL). Analysis was performed on per protocol set. Only participants with data available at specified timepoint were included in the analysis.
Time Frame: At Day 43
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | MMRV(H)NS Vaccine | MM(H)RVNS Vaccine | (MMRV)(L)NS Vaccine | MMRV_Lot 1 and Lot 2 Pooled Group
Number analyzed (Participants) | 167 | 171 | 162 | 168
IU/mL | 159 (145) [145 to 173] | 178 (163) [163 to 195] | 158 (144) [144 to 172] | 149 (137) [137 to 163]

4. Primary Outcome: GMC of Anti-glycoprotein E (gE) Antibodies at Day 43
Description: Anti-gE antibodies were measured with enzyme linked immunosorbent assay and the results were expressed as GMC, in mIU/mL. Anti-varicella and anti-varicella zoster virus gE were used interchangeably. Analysis was performed on per protocol set. Only participants with data available at specified timepoint were included in the analysis.
Time Frame: At Day 43
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | MMRV(H)NS Vaccine | MM(H)RVNS Vaccine | (MMRV)(L)NS Vaccine | MMRV_Lot 1 and Lot 2 Pooled Group
Number analyzed (Participants) | 170 | 172 | 165 | 169
mIU/mL | 4229 (3723) [3723 to 4804] | 3743 (3257) [3257 to 4303] | 3369 (2934) [2934 to 3867] | 4002 (3493) [3493 to 4585]

5. Secondary Outcome: Percentage of Participants With Seroresponse for Measles Antibodies at Day 43
Description: Seroresponse was defined as the participants of participants for whom the Day 43 measles antibodies concentration was >=116 mIU/mL. Analysis was performed on per protocol set. Only participants with data available at specified timepoint were included in the analysis.
Time Frame: At Day 43
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MMRV(H)NS Vaccine | MM(H)RVNS Vaccine | (MMRV)(L)NS Vaccine | MMRV_Lot 1 and Lot 2 Pooled Group
Number analyzed (Participants) | 167 | 171 | 162 | 168
Percentage of participants | 99.4 (96.71) [96.71 to 99.98] | 98.2 (94.96) [94.96 to 99.64] | 96.3 (92.11) [92.11 to 98.63] | 95.2 (90.83) [90.83 to 97.92]

6. Secondary Outcome: Percentage of Participants With Seroresponse for Mumps Antibodies at Day 43
Description: Seroresponse was defined as the participants of participants for whom the Day 43 mumps antibodies concentration was >=296 AU/mL. Analysis was performed on per protocol set. Only participants with data available at specified timepoint were included in the analysis.
Time Frame: At Day 43
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MMRV(H)NS Vaccine | MM(H)RVNS Vaccine | (MMRV)(L)NS Vaccine | MMRV_Lot 1 and Lot 2 Pooled Group
Number analyzed (Participants) | 167 | 171 | 162 | 168
Percentage of participants | 98.8 (95.74) [95.74 to 99.85] | 100.0 (97.87) [97.87 to 100.0] | 100.0 (97.75) [97.75 to 100.0] | 99.4 (96.73) [96.73 to 99.98]

7. Secondary Outcome: Percentage of Participants With Seroresponse for Rubella Antibodies at Day 43
Description: Seroresponse was defined as the participants of participants for whom the Day 43 rubella antibodies concentration was >=24 IU/mL. Analysis was performed on per protocol set. Only participants with data available at specified timepoint were included in the analysis.
Time Frame: At Day 43
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MMRV(H)NS Vaccine | MM(H)RVNS Vaccine | (MMRV)(L)NS Vaccine | MMRV_Lot 1 and Lot 2 Pooled Group
Number analyzed (Participants) | 167 | 171 | 162 | 168
Percentage of participants | 100.0 (97.82) [97.82 to 100.0] | 100.0 (97.87) [97.87 to 100.0] | 100.0 (97.75) [97.75 to 100.0] | 100.0 (97.83) [97.83 to 100.0]

8. Secondary Outcome: Percentage of Participants With Seroresponse for Varicella Antibodies at Day 43
Description: Seroresponse was defined as the participants of participants for whom the Day 43 varicella antibodies concentration was >=300 mIU/mL. Analysis was performed on per protocol set. Only participants with data available at specified timepoint were included in the analysis.
Time Frame: At Day 43
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MMRV(H)NS Vaccine | MM(H)RVNS Vaccine | (MMRV)(L)NS Vaccine | MMRV_Lot 1 and Lot 2 Pooled Group
Number analyzed (Participants) | 170 | 172 | 165 | 169
Percentage of participants | 100.0 (97.85) [97.85 to 100.0] | 100.0 (97.88) [97.88 to 100.0] | 100.0 (97.79) [97.79 to 100.0] | 100.0 (97.84) [97.84 to 100.0]

9. Secondary Outcome: Number of Participants With Solicited Administration Site Adverse Events (AEs) During the 4-day Period After Vaccine Dose Administration
Description: The solicited administration site events after vaccination included pain, erythema/redness, and swelling. Analysis was performed on exposed set which included all participants who received a study intervention. Only those participants with solicited AEs were included in this analysis.
Time Frame: Day 1 to Day 4
Measure: Count of Participants; unit: Participants
Arm/Group | MMRV(H)NS Vaccine | MM(H)RVNS Vaccine | (MMRV)(L)NS Vaccine | MMRV_Lot 1 and Lot 2 Pooled Group
Number analyzed (Participants) | 198 | 200 | 203 | 195
Participants
  Injection site pain | 76 | 58 | 64 | 76
  Redness at injection site | 41 | 34 | 26 | 42
  Swelling at injection site | 24 | 21 | 14 | 20

10. Secondary Outcome: Number of Participants With Solicited Systemic AEs During the 4-day Period After Vaccine Dose Administration
Description: The solicited systemic events after vaccination included drowsiness and loss of appetite. Analysis was performed on exposed set. Only those participants with solicited AEs were included in this analysis.
Time Frame: Day 1 to Day 4
Measure: Count of Participants; unit: Participants
Arm/Group | MMRV(H)NS Vaccine | MM(H)RVNS Vaccine | (MMRV)(L)NS Vaccine | MMRV_Lot 1 and Lot 2 Pooled Group
Number analyzed (Participants) | 198 | 200 | 203 | 195
Participants
  Any drowsiness | 27 | 18 | 32 | 31
  Any loss of appetite | 20 | 14 | 22 | 26

11. Secondary Outcome: Number of Participants With Solicited Systemic AEs During the 43-day Period After Vaccine Dose Administration
Description: The solicited systemic events after vaccination included fever, measles/rubella-like rash, varicella- like rash and other rash (not measles/rubella-like rash or varicella-like rash). Fever was defined as temperature greater than or equal to 38.0 degrees Celsius (100.4 degrees Fahrenheit) by any route (the preferred location for measuring temperature is the axilla). Analysis was performed on exposed set. Only those participants with solicited AEs were included in this analysis.
Time Frame: Day 1 to Day 43
Measure: Count of Participants; unit: Participants
Arm/Group | MMRV(H)NS Vaccine | MM(H)RVNS Vaccine | (MMRV)(L)NS Vaccine | MMRV_Lot 1 and Lot 2 Pooled Group
Number analyzed (Participants) | 198 | 200 | 203 | 195
Participants
  Fever | 27 | 25 | 25 | 27
  Any measles/rubella-like rash | 13 | 8 | 12 | 5
  Any varicella-like rash (including injection site) | 5 | 6 | 6 | 6
  Any other rash | 16 | 18 | 19 | 14

12. Secondary Outcome: Number of Participants With Unsolicited AEs During the 43-day Period After Vaccine Dose Administration
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study vaccine, which does not necessarily have a causal relationship with study vaccine. An unsolicited AE was an AE that was either not included in the list of solicited events or was included in the list of solicited events but with an onset outside the specified period of follow- up for solicited events. Unsolicited AEs must have been communicated by participant/participant's caregiver(s) who had signed the informed consent. Unsolicited AEs included both serious adverse events (SAEs) and non-serious AEs. Analysis was performed on exposed set.
Time Frame: Day 1 to Day 43
Measure: Count of Participants; unit: Participants
Arm/Group | MMRV(H)NS Vaccine | MM(H)RVNS Vaccine | (MMRV)(L)NS Vaccine | MMRV_Lot 1 and Lot 2 Pooled Group
Number analyzed (Participants) | 198 | 200 | 203 | 195
Participants | 44 | 37 | 48 | 53

13. Secondary Outcome: Number of Participants With SAEs After Vaccine Dose Administration
Description: An SAE was defined as any untoward medical occurrence that, at any dose, resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, resulted in congenital anomaly or other significant medical events. Analysis was performed on exposed set.
Time Frame: Throughout the study period (Day 1 to Day 181)
Measure: Count of Participants; unit: Participants
Arm/Group | MMRV(H)NS Vaccine | MM(H)RVNS Vaccine | (MMRV)(L)NS Vaccine | MMRV_Lot 1 and Lot 2 Pooled Group
Number analyzed (Participants) | 198 | 200 | 203 | 195
Participants | 1 | 1 | 1 | 1

ADVERSE EVENTS:
Time Frame: Solicited administration site and systemic events (drowsiness, loss of appetite): Day 1 to 4; solicited systemic events (fever, measles/rubella like rash, varicella-like rash and other rash); and unsolicited AEs: Day 1 to 43; SAEs: Day 1 to 181
Description: Solicited and unsolicited events were reported per participant/parent at any dose for the assessed timeframe (within 43 days after vaccine dose administration) according to occurrence of each event, as pre-specified in Statistical Analysis Plan.
Arm/Group | MMRV(H)NS Vaccine | MM(H)RVNS Vaccine | (MMRV)(L)NS Vaccine | MMRV_Lot 1 and Lot 2 Pooled Group
All-Cause Mortality (participants affected / at risk) | 1/198 | 0/200 | 0/203 | 0/195
Serious Adverse Events (participants affected / at risk) | 1/198 | 1/200 | 1/203 | 1/195
Other Adverse Events (participants affected / at risk) | 127/198 | 114/200 | 126/203 | 132/195
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MMRV(H)NS Vaccine (N=198) | MM(H)RVNS Vaccine (N=200) | (MMRV)(L)NS Vaccine (N=203) | MMRV_Lot 1 and Lot 2 Pooled Group (N=195)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Homicide (Social circumstances) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MMRV(H)NS Vaccine (N=198) | MM(H)RVNS Vaccine (N=200) | (MMRV)(L)NS Vaccine (N=203) | MMRV_Lot 1 and Lot 2 Pooled Group (N=195)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal pruritus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Salivary gland enlargement (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2) | 3 (3)
Administration site erythema (General disorders) | 41 (71) | 34 (62) | 26 (50) | 42 (63)
Administration site pain (General disorders) | 76 (114) | 58 (76) | 64 (89) | 76 (108)
Administration site swelling (General disorders) | 24 (35) | 21 (35) | 14 (22) | 20 (27)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 4 (4) | 3 (3) | 0 (0) | 3 (3)
Injection site induration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 2 (2) | 4 (4) | 4 (4) | 3 (3)
Injection site swelling (General disorders) | 3 (3) | 3 (3) | 0 (0) | 1 (1)
Injection site urticaria (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site warmth (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 27 (45) | 25 (60) | 25 (49) | 27 (52)
Seasonal allergy (Immune system disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Croup infectious (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Herpangina (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2) | 5 (6) | 5 (5)
Otitis media (Infections and infestations) | 4 (4) | 2 (2) | 3 (3) | 1 (1)
Otitis media acute (Infections and infestations) | 4 (4) | 1 (1) | 2 (2) | 3 (3)
Pharyngitis (Infections and infestations) | 2 (2) | 2 (2) | 3 (3) | 2 (2)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pustule (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scarlet fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin candida (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinea capitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 9 (9) | 7 (8) | 7 (7) | 10 (10)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Viral pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctival abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Abnormal weight gain (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 20 (24) | 14 (20) | 22 (26) | 26 (33)
Overweight (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 27 (34) | 18 (33) | 32 (39) | 32 (46)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Autism spectrum disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Behavioural insomnia of childhood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oppositional defiant disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tic (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urethral meatus stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 1 (1) | 5 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rashes, eruptions and exanthems NEC (Skin and subcutaneous tissue disorders) | 24 (112) | 23 (128) | 27 (113) | 17 (108)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT05630846/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-11): https://cdn.clinicaltrials.gov/large-docs/46/NCT05630846/SAP_001.pdf